CLINICAL TRIAL: NCT06499623
Title: Early Detection of Malnutrition in Oncology Patients and People Over 65 Years of Age
Brief Title: Early Detection of Malnutrition in Oncology Patients and Elderly Patients
Acronym: MALNUTRITION
Status: Recruiting | Type: Observational
Sponsor: Institute of Health Information and Statistics of the Czech Republic (Other Government)
Collaborators: Brno University Hospital (Other); Bulovka Hospital (Other); Masaryk Memorial Cancer Institute (Other); University Hospital, Motol (Other); Hospital AGEL Nový Jičín a.s. (Unknown); Military University Hospital, Prague (Other); General University Hospital, Prague (Other); University Hospital Olomouc (Other); University Hospital Pilsen (Other)
Responsible Party: Sponsor
Other Study IDs: UZIS 2024/1
Record Dates: First submitted 2024-07-08; First posted 2024-07-12 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Malnutrition
Keywords: malnutrition; oncology; gerontology
MeSH Terms: conditions — Malnutrition; Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Oncological patients: The inclusion criteria for the cohort of oncological patients are age 18+, an oncological diagnosis and a survival prognosis of at least 3 months.
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Bioelectrical Impedance Analysis; Other: Nutritional Risk Assessment Questionnaire
- Patients older than 65 years: The inclusion criteria for this cohort are age 65 and older and hospitalization at least 14 days or longer.
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Bioelectrical Impedance Analysis; Other: Nutritional Risk Assessment Questionnaire

INTERVENTIONS:
Diagnostic Test: Blood test — Albumin, C-Reactive Protein, Cholesterol, Urea, Creatinine, Vitamin D
Diagnostic Test: Bioelectrical Impedance Analysis — Total Impedance, Segmental Muscle Analysis, Segmental Fat Analysis, Absolute Muscle Mass Value, Muscle Mass Index, Total Body Fat Percentage, Total Body Water, Phase Angle Measurement
Other: Nutritional Risk Assessment Questionnaire — Fill in the Questionnaire of the Working Group on Nutritional Care in Oncology and get nutrition risk score. The objective data includes weight loss in 6 months, current BMI and food tolerance, and oncological diagnosis including ongoing anti-cancer treatment.

SUMMARY:
The project is a national, prospective, multicenter, non-interventional pilot project of malnutrition screening in the Czech Republic.

The main goal of the project is to methodically prepare, implement and evaluate a pilot project that will verify the suitability of the proposed procedure for the early detection of malnutrition in oncology patients and hospitalised patients patients 65 years of age and older, as this has a significant effect on the quality of life and the effectiveness of the services provided oncological treatment.

DETAILED DESCRIPTION:
The main goal of the project is the early detection of malnutrition in oncology patients and hospitalised patients 65 years of age and older, as this has a significant effect on the quality of life and the effectiveness of the services provided oncological treatment.

Another goal of the project will be the creation of a unified diagnostic proposal process and methodological material for determining malnutrition. This process will then be designed as the standard of nursing practice for patients with an oncological diagnosis and for persons older than 65 years such that, so that an adequate nutritional intervention is started in time, which will lead to a higher tolerance of demanding treatment and thus to increase the quality of life.

The project will include testing the procedure on a sample of approx. 1,500 oncological and 500 geriatric patients.

The project is supported by the European Social Fund (Operational Program Employment plus) and the state budget of the Czech Republic and is registered by the Ministry of Labour and Social Affairs of the Czech Republic under ID: CZ.03.02.02/00/22_005/0000282.

ELIGIBILITY:
Inclusion Criteria:

Cohort Oncological patients:

* 18+
* an oncological diagnosis
* a survival prognosis of at least 3 months

Cohort Patients older than 65 years:

* 65+
* hospitalization at least 14 days or longer

Exclusion Criteria (both cohorts):

* not agreeing to participate in the project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with oncological diagnosis with age 18+ or patients with hospitalization at least 14 days and age 65+.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of people with malnutrition according to the PSNPO questionnaire | Until 31. 3. 2026

SECONDARY OUTCOMES:
Proportion of people with initiated nutritional intervention | Until 31. 3. 2026

CONTACTS AND LOCATIONS:
Overall Officials: Petra Beran Holeckova, MD, Study Director — Charles University First Faculty of Medicine
Locations (9):
- Czechia (9):
  - Brno University Hospital, Brno
  - Masaryk Memorial Cancer Institute, Brno
  - Hospital AGEL Nový Jičín a.s., Nový Jičín
  - University Hospital Olomouc, Olomouc
  - University Hospital Pilsen, Pilsen
  - Bulovka Hospital, Prague
  - General University Hospital, Prague, Prague
  - Military University Hospital, Prague, Prague
  - University Hospital, Motol, Prague

IPD SHARING:
Plan to Share IPD: No